CLINICAL TRIAL: NCT04020523
Title: Evaluation of Advanced MRI Acquisition Techniques for Perfusion and Diffusion to Detect Breast Cancer
Brief Title: Advanced MR Techniques for Breast Cancer Detection
Acronym: RAPIDIRM
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Delayed start due to technical problems as well as the covid pandemic. Decision of the investigator
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: K180603J; 2018-A01647-48 (Other: ANSM)
Record Dates: First submitted 2019-05-24; First posted 2019-07-16 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Breast Cancer
Keywords: MRI; breast; cancer; screening; innovative sequences
MeSH Terms: conditions — Breast Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient with an injected breast MR exam (Experimental)
  Interventions: Other: MRI sequence

INTERVENTIONS:
Other: MRI sequence — The MR sequences added to the protocol are dedicated sequences for perfusion and diffusion imaging of breast lesion.

SUMMARY:
Evaluation of advanced MRI acquisition techniques (perfusion and diffusion) to detect breast cancer. Two MR advanced sequences will be added to a standard breast MRI protocol for evaluation purpose.

DETAILED DESCRIPTION:
This is a prospective monocentric longitudinal study on a consecutive population of patients who require breast MRI as part of their course of care in the radiology department of the Tenon Hospital (3T MRI).

The standard protocol for breast MRI routinely performed in Tenon hospital consists of a set of MR acquisitions performed with contrast agent injection. The research consists of adding perfusion and diffusion sequences to the regular MR protocol. The addition of these sequences does not require a new injection of contrast medium.

Diagnosis of lesions after the breast MR exam will be performed using standard MR sequences as usual. According to the recommendations of SIFEM, the final diagnosis of the lesions will be made either by histological analysis of a biopsy performed as part of the patient's standard care pathway, or during patient's follow-up if a biopsy is not indicated (up to two years after breast MR exam).

The research will focus on evaluating the sensitivity and specificity of perfusion MRI sequence with or without diffusion MRI sequence compared to the sensitivity and specificity of the standard protocol.

For the perfusion sequence, the following data will be extracted: qualitative (shape of the contrast curve), semi-quantitative (elevation slope and asymptote of the curve) and quantitative by compartmental modeling (tissue perfusion, blood volume fraction, surface capillary permeability).

For the diffusion MRI, the extraction of quantitative data such as CDA, IVIM and Kurtosis will be performed and parametric maps, cellularity maps and an assessment of lesion heterogeneity will be calculated.

A correlation will be made with histological, immunohistochemical and molecular results of cancers following biopsy

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Patient who has signed a consent form to participate in the study
* Affiliated patient or beneficiary of a social security scheme
* Patient with an injected breast MR exam planned as part of her care pathway.

Exclusion Criteria:

* Patients under guardianship or curatorship
* Pregnant or breastfeeding patients
* Patients with contraindications to realization of an MR exam and an injected MR exam

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-07 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Mammary lesions Visualization on ultrafast injected dynamic MRI: Yes/No | Day 1 at inclusion
  to evaluate whether ultrafast injected dynamic breast MRI, coupled or not with a diffusion sequence, allows to improve the specificity of standard MRI while maintaining the same sensitivity
Mammary lesions Visualization with a diffusion sequence | Day 1 at inclusion
  to evaluate whether ultrafast injected dynamic breast MRI, coupled or not with a diffusion sequence, allows to improve the specificity of standard MRI while maintaining the same sensitivity

SECONDARY OUTCOMES:
Quantitative perfusion parameters : Enhancement Integral (EI (%)) | Day 1 at inclusion
  Correlate the parameters of perfusion MR sequence with the markers immunochemicals of tumor angiogenesis on anatomopathological specimen
Quantitative perfusion parameters : Maximum Slope of Increase (MSI (%/sec)) | Day 1 at inclusion
  Correlate the parameters of perfusion MR sequence with the markers immunochemicals of tumor angiogenesis on anatomopathological specimen
Quantitative perfusion parameters : Maximum of enhancement (Rmax (%)) | Day 1 at inclusion
  Correlate the parameters of perfusion MR sequence with the markers immunochemicals of tumor angiogenesis on anatomopathological specimen
Quantitative perfusion parameters : Timing of Maximum of enhancement (RmaxTiming (sec)) | Day 1 at inclusion
  Correlate the parameters of perfusion MR sequence with the markers immunochemicals of tumor angiogenesis on anatomopathological specimen
Quantitative perfusion parameters : Wash-inrate (WIR (%/sec) | Day 1 at inclusion
  Correlate the parameters of perfusion MR sequence with the markers immunochemicals of tumor angiogenesis on anatomopathological specimen
Correlate diffusion MRI parameters with immunochemical markers of tumor angiogenesis on anatomopathological specimen Quantitative diffusion parameter : Apparent Coefficient Diffusion | Day 1 at inclusion
Evaluate the reduction in the time required to acquire and interpret the new breast MR protocol compared to the standard one | Day 1 at inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle THOMASSIN-NAGGARA, PU-PH, Principal Investigator — Assistance Publique - Hôpitaux de Paris